CLINICAL TRIAL: NCT06843577
Title: A Pivotal Study to Evaluate the Effectiveness of Isometric Handgrip Therapy in Elevated Blood Pressure and Hypertensive Subjects
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zona Health, Inc (Industry)
Collaborators: Emergent Clinical Consulting, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Zona-002
Record Dates: First submitted 2025-02-20; First posted 2025-02-25 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Elevated Blood Pressure; Hypertension
Keywords: Hypertension; Elevated Blood Pressure
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Investigational (Experimental): Zona Plus Device
- Control (Active Comparator): Relaxing music
  Interventions: Other: Relaxing Music App

INTERVENTIONS:
Device: Zona Plus Device — Use of the Zona Plus device involves performing isometric handgrip exercise therapy. Isometric exercise is the type of exercise in which you tense or tighten your muscle without seeing it change in length.
Other: Relaxing Music App — Relaxing music will be made available through a mobile app that users access via their smart phone or tablet. Subjects will have the option to listen to 5 different music genres that support relaxation (Classical, Nature, Movie Soundtracks, Jazz, Reggae).
  Arms: Control

SUMMARY:
The study will be a multi-center, randomized clinical trial to evaluate the safety and efficacy of using the Zona Plus handgrip therapy device compared to the use of an auditory relaxation therapy for treatment of high blood pressure and hypertension in subjects who are not currently taking antihypertensive medications. Half of the study subjects will also be randomized to record blood pressure at home throughout the study.

DETAILED DESCRIPTION:
Study subjects randomized to the Zona Plus Device arm will perform isometric therapy with the device with subject compliance monitored through a downloadable electronic memory function built into the device. Study subjects randomized to the control arm will be asked to listen to relaxing music via a mobile app and asked to document their compliance via a patient diary. Subjects in the control arm may be able to crossover to using the Zona Plus device after completion of Study Visit 6. Subjects who have systolic blood pressure between 140mmHG and 149mmHG at baseline will complete three additional study visits for further monitoring. Subjects can expect participation in the study to last between 3 and 8 months.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is male or female age 22 or older
2. Diagnosed with elevated blood pressure or hypertension and verified during Visit #1 by standardized seated cuff SBP
3. Have not taken antihypertensive medication for ≥30 days prior to the SEPV
4. Subject is expected to have sufficient vision, hearing, and hand strength (hand strength is demonstrated by a maximum voluntary contraction (MVC) equaling 35 units of force in both hands measured by a dynamometer
5. Subject has baseline BP measurements collected and completes study device training during Baseline Assessment (Visit #1);
6. Subject agrees to maintain non-use of medications and over-the-counter (OTC) supplement regimen related to hypertension throughout the treatment phase;
7. Patient can comply with and agrees to complete all required study procedures, study clinic visits, and associated activities;
8. Patient must be able to understand and give written informed consent in the language provided;
9. Subject must have SBP of 130 to ≤149 mmHg, if subjects present with SBP reading of ≥140mmHg they will receive heightened monitoring throughout the first month of the study

Exclusion Criteria:

1. Subject is a female of childbearing potential (e.g., not postmenopausal for at least one year or has not had a hysterectomy or tubal ligation) not using medically effective birth control (e.g., hormonal methods in use at least 30 days prior to screening or barrier methods such as condom and spermicide in use at least 14 days prior to visit 1) or is pregnant, lactating, or plans to become pregnant during the study).
2. BP ≥150 mmHg (systolic) and/or >90 mmHg (diastolic)
3. A history of heart failure with current New York Heart Association (NYHA) class III- IV functional classification
4. Currently has, or has had a history, of atrial fibrillation, in accordance with 2007 Heart Rhythm Society (HRS)/European Heart Rhythm Association (EHRA)/European Cardiac Arrhythmia Society (ECAS) guidelines
5. Patient has experienced hospitalization due to a hypertensive emergency, with impending or progressive target organ dysfunction (i.e., renal dysfunction, left ventricular hypertrophy or CNS involvement) within the past six (6) months
6. A >10 mmHg difference in seated cuff SBP between the right and left arms collected during the SEPV;
7. Unstable BP, defined as >5 mmHg variance between any two (2) consecutive weekly readings (with a maximum of four (4) attempts) to determine a baseline BP measurement ;
8. Arm circumference greater than 45 cm;
9. Acute illness, infection, or inflammation
10. Presence of any unstable cardiovascular disorder, such as MI, unstable angina, significant arrhythmia, stroke, or TIA; within the last six (6) months, or other serious comorbidity that would be likely to impact life expectancy to less than one (1) year or limit patient cooperation or study compliance;
11. A history of rest or exertional angina pectoris in the previous six (6) months;
12. History of solid organ transplant
13. Any secondary form of hypertension (HTN) etiology, including but not limited to primary aldosteronism, chronic steroid therapy and Cushing syndrome, pheochromocytoma, aorta coarctation or untreated thyroid or parathyroid disease;
14. Concurrent participation in an investigational clinical study that has not completed the follow-up period or planned participation in another study within the next six (6) months;
15. Patient has any other condition or personal circumstance that, in the judgment of the investigator, might interfere with the collection of complete, good quality data or the completion of the research study;
16. Patients who currently own or have owned another Zona Plus device and are, or have been, voluntarily performing the isometric handgrip activities.
17. Subject plans for greater than 10% of body weight loss/gain (10% of body weight over a 6-month period) during the study

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-03-27 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Compare the change from baseline in mean seated cuff systolic blood pressure (SBP) after 10 weeks of treatment between patients randomized to the Zona Plus device and the patients in the control group. | 10 weeks

SECONDARY OUTCOMES:
To compare the change from baseline in seated cuff diastolic blood pressure ("DBP") after 10 weeks of treatment between patients randomized to the Zona Plus device and the patients in the control group. | 10 weeks
The percentage of patients randomized to the Zona Plus device who achieve a clinically significant SBP reduction (defined as ≥5 mmHg) at Week 10 compared to control. | 10 weeks
The percentage of patients randomized to the Zona Plus device who achieve a clinically significant DBP reduction (defined as ≥3 mmHg) at Week 10 compared to control. | 10 weeks

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Bayview Research Group, Valley Village, California
  - AMR Miami, Coral Gables, Florida
  - Cedar Crosse Research Center, Chicago, Illinois
  - Circuit Clinical Grave Gilbert, Bowling Green, Kentucky
  - AMR Knoxville, Knoxville, Tennessee

IPD SHARING:
Plan to Share IPD: No